CLINICAL TRIAL: NCT02388464
Title: A Phase 1 Clinical Pharmacology Study of the Effects of a Single 4 Hour Intravenous Infusion of Bendavia™ (MTP-131) in Subjects With Stable New York Heart Association Class II-III Congestive Heart Failure Due to Left Ventricular Systolic Dysfunction
Brief Title: A Study Investigating the Safety, Tolerability, and Pharmacokinetics of MTP-131 in Subjects With Congestive Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPIHF-101
Record Dates: First submitted 2015-03-01; First posted 2015-03-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Bendavia™; MTP-131
MeSH Terms: conditions — Heart Failure | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose (Experimental)
  Interventions: Drug: MTP-131
- Intermediate dose (Experimental)
  Interventions: Drug: MTP-131
- High dose (Experimental)
  Interventions: Drug: MTP-131
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MTP-131 — MTP-131 (low dose) administered as single intravenous infusion over 4 hours
  Arms: Low dose
Drug: MTP-131 — MTP-131 (intermediate dose) administered as single intravenous infusion over 4 hours
  Arms: Intermediate dose
Drug: MTP-131 — MTP-131 (high dose) administered as single intravenous infusion over 4 hours
  Arms: High dose
Drug: Placebo — Placebo Comparator (at each dose cohort) administered as single intravenous infusion over 4 hours
  Arms: Placebo

SUMMARY:
This is a Phase 1, single-center, randomized, double-blind, single ascending dose, placebo-controlled study, in subjects aged 45-80 years with stable mild to moderate heart failure due to left ventricular systolic dysfunction, to evaluate the safety, tolerability, and pharmacokinetics of escalating single intravenous infusion doses of Bendavia™ (MTP-131).

ELIGIBILITY:
Inclusion Criteria:

* Chronic ischemic or non-ischemic cardiomyopathy of at least 6 months duration from the time of the initial diagnosis.
* LVEF ≤35% by 2-D echocardiogram.
* Diagnosis of NYHA Class II or III HF for a minimum of 6 months prior to the Screening Visit.
* HF is considered to be stable and no hospitalization for HF has occurred within the previous 3 months prior to the Screening visit.
* Treatment with appropriate pharmacologic therapy for HF including, but not limited to, angiotensin converting enzyme inhibitor (ACEI) and/or angiotensin receptor blocker (ARB), and an evidence-based beta blocker for the treatment of HF (i.e. carvedilol, bisoprolol, or extended-release metoprolol).
* Dose and dose regimen of pharmacologic treatments for HF must be stable for a minimum of 1 month prior to the Screening Visit.
* Females of child-bearing potential must have a negative serum pregnancy test at the Screening Visit and Day 1.

Exclusion Criteria:

* LV end-diastolic dimension (LVEDD), by the same method as qualifying LVEF, is >80 mm or LVEDD indexed to body surface area is >0.45.
* Unstable angina pectoris within 1 month before initiation of screening procedures. Unstable angina is defined as the occurrence of chest pain more frequently than usual, pain at rest or upon minimal exertion, or protracted episodes of pain without any discernible trigger, and/or chest pain that persists despite use of vasodilatory therapy (e.g., nitroglycerin).
* Coronary or peripheral artery revascularization procedure within 2 months prior to the Screening Visit.
* An acute myocardial infarction within 3 months prior to the Screening Visit.
* Placement of an automated implantable cardioverter defibrillator (AICD) or any hardware associated with resynchronization therapy.
* Atrial fibrillation at the Screening or Baseline Visits.
* Uncontrolled hypertension defined as a systolic blood pressure (BP) > 180 mm Hg or a diastolic BP >110 mm Hg on at least 2 consecutive readings.
* Requirement for valve or other cardiac surgery
* Cardiac surgery or valvuloplasty within 2 months prior to the Screening Visit.
* General surgery within 1 month prior to the Screening Visit
* Restrictive cardiomyopathy, obstructive cardiomyopathy, pericardial disease, amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease, or dyskinetic left ventricular aneurysm.
* Cerebrovascular accident or transient ischemic attack within 3 months prior to the Screening Visit.
* Estimated glomerular filtration rate (eGFR) <40 mL/min, using the Modification of Diet in Renal Disease (MDRD) Study equation
* Serologic evidence of hepatitis B or C infection.
* Known acquired immunodeficiency syndrome or HIV-positive status, or diagnosis of immunodeficiency.

  * Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Assessed up to Day 7

SECONDARY OUTCOMES:
Left ventricular ejection fraction assessed by 2-D echocardiography | Assessed up to 24 hours post-infusion start

CONTACTS AND LOCATIONS:
Overall Officials: Jim Carr, PharmD, Study Director — Stealth BioTherapeutics Inc.; Sotir Marchev, MD,PhD, FESC, Principal Investigator — Bulgaria
Locations (1):
- Sevlievo, Gabrovo, Bulgaria

REFERENCES:
- [Derived] Daubert MA, Yow E, Dunn G, Marchev S, Barnhart H, Douglas PS, O'Connor C, Goldstein S, Udelson JE, Sabbah HN. Novel Mitochondria-Targeting Peptide in Heart Failure Treatment: A Randomized, Placebo-Controlled Trial of Elamipretide. Circ Heart Fail. 2017 Dec;10(12):e004389. doi: 10.1161/CIRCHEARTFAILURE.117.004389. PMID 29217757